CLINICAL TRIAL: NCT02199821
Title: Inflammatory Response With Different Lipid Emulsions In Parenteral Nutrition In Children After Bone Marrow Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PI-00000
Record Dates: First submitted 2014-04-30; First posted 2014-07-25 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-05

CONDITIONS: Bone Narrow Transplantation
MeSH Terms: interventions — Food, Formulated; Soybean Oil

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Soybean oil formula commonly used in the hospita (Active Comparator)
  Interventions: Dietary Supplement: Soybean oil formula commonly used in the hospital
- Formula with soybean oil, medium-chain triglyce (Experimental)
  Interventions: Dietary Supplement: Formula with soybean oil, medium-chain triglycerides

INTERVENTIONS:
Dietary Supplement: Formula with soybean oil, medium-chain triglycerides
  Arms: Formula with soybean oil, medium-chain triglyce
Dietary Supplement: Soybean oil formula commonly used in the hospital
  Arms: Soybean oil formula commonly used in the hospita

SUMMARY:
Background and Aims: Nutritional support is considered an integral part of the supportive care of bone marrow transplantation patients. Parenteral nutrition emulsions enriched with omega-3 fatty acids can modify the inflammatory response. The aim of this study is to compare plasma cytokines levels in children after bone marrow transplantation using a lipid formula enriched in n-3 FA and other classic soybean oil formula in parenteral nutrition.

Methods: A randomized double blinded controlled study including 14 children with BMT and requiring PN for at least 10 days was conducted using a lipid emulsion with fish oil, or soybean oil. Blood samples at baseline, at 10 days and at the end of the PN were taken to analyze plasma interleukins 1 beta, 2, 6, 8, 10 (IL-10) and tumor necrosis factor alpha (TNF-α).

ELIGIBILITY:
Inclusion Criteria:

Term infants. Children with a stable medical condition. Children in need of parenteral nutrition for at least 10 days, except for the cardiac group would be at least 5 days.

Exclusion Criteria:

Premature infants Children over 14 years Children with hypersensitivity to egg ingestion or soy protein Children with severe insufficiency of an organ, Children with inborn error of metabolism, and any condition that does not allow random use of lipid emulsion type.

Ages: 1 Day to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2011-02; Primary Completion 2013-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
average cytokines plasma levels between groups of children with the two different lipid formulas. | 21 days
  The primary outcome of the trial was average cytokines plasma levels between groups of children with the two different lipid formulas.

SECONDARY OUTCOMES:
Anthropometric measurements such as: weight height | 21 days
Incidence of adverse effects associated with formula consumption. | 21 days